CLINICAL TRIAL: NCT06278675
Title: A Multicenter Clinical Study on the Effect of Electroacupuncture on the Mechanical Ventilation Strategy in Patients With Sepsis-related ARDS
Brief Title: Multiple Study of Electroaccpuncture in ARDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jun Lu, MD, Director, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEOVA
Record Dates: First submitted 2024-02-12; First posted 2024-02-26 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acute Respiratory Distress Syndrome; Sepsis
MeSH Terms: conditions — Respiratory Distress Syndrome; Sepsis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group: Sterile stainless steel needle electroacupuncture treatment was applied, and the acupuncture points were as follows: bilateral Zusanli (ST36), Neiguan (PC6), Hegu (LI4), Shaoshang (LU11), and Feng Long (ST40). 1 time a day, 30 minutes each time, for 7 days.
  Interventions: Device: Acupuncture needles
- Control group (No Intervention): Control group: Placebo needles were applied, and the acupuncture points were as follows: bilateral Zusanli (ST36), Neiguan (PC6), Hegu (LI4), Shaoshang (LU11), and Feng Long (ST40). 1 time a day, 30 minutes each time, for 7 days.

INTERVENTIONS:
Device: Acupuncture needles — 1. Experimental group: Sterile stainless steel needle electroacupuncture treatment was applied, and the acupuncture points were as follows: bilateral Zusanli (ST36), Neiguan (PC6), Hegu (LI4), Shaoshang (LU11), and Feng Long (ST40). 1 time a day, 30 minutes each time, for 7 days.
  2. Control group: Placebo needles were applied, and the acupuncture points were as follows: bilateral Zusanli (ST36), Neiguan (PC6), Hegu (LI4), Shaoshang (LU11), and Feng Long (ST40). 1 time a day, 30 minutes each time, for 7 days.
  Arms: Experimental group

SUMMARY:
In order to clarify the clinical efficacy of electroacupuncture on inhibiting systemic inflammatory response, improving respiratory mechanics parameters and prognosis in patients with sepsis-related ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of the Surviving Sepsis Campaign: Updated International Guidelines for the Treatment of Sepsis and Septic Shock 2021
* Meet the diagnostic criteria of the European Society of Critical Care Medicine (ESICM) Guidelines for Acute Respiratory Distress Syndrome: Definition, Phenotype and Respiratory Support Strategies
* Age >18 years
* Expected duration of mechanical ventilation>48 hours
* Expected ICU stay of more than 7 days
* Signed informed consent.

Exclusion Criteria:

* Participated in other clinical trials
* Pregnant, lactating or miscarriage
* Patients with disseminated tumors or tumors receiving chemotherapy and other special treatments
* Alcohol abuse
* Severe cardiovascular, brain, liver, kidney, psychiatric diseases, diabetes, multiple system atrophy, cauda equina injury or myelopathy
* Systolic blood pressure < 90mmHg within 2 hours before the start of the study
* Severe burns or severe skin diseases
* Pacemaker placement, metal allergy or severe needle sickness
* Abnormal coagulation function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory mechanics indicators 1 | Day 0、day 7
  Oxygenation index(P/F)
Respiratory mechanics indicators 2 | Day 0、day 7
  Respiratory rate(RR)
Respiratory mechanics indicators 3 | Day 0、day 7
  Driving pressure(DP)
Respiratory mechanics indicators 4 | Day 0、day 7
  Positive end expiratory pressure(PEEP)
Respiratory mechanics indicators 5 | Day 0、day 7
  Mechanical ventilation days(MV days)
Respiratory mechanics indicators 6 | Day 0、day 7
  Mechanical ventilation free days(MV free days)
Respiratory mechanics indicators 7 | Day 0、day 7
  Extubation situation

SECONDARY OUTCOMES:
Sedation and analgesia | Day 0、day 7
  RASS score
Sedative drug use | Day 0、day 7
  The dose and duration of sedative medication will be recorded.
Analgesic drug use | Day 0、day 7
  The dose and duration of analgesic medication will be recorded.
Inflammatory factors | Day 0、day 7
  IL-1β、IL-6、IL-2、IL-4、IL-5、IL-8、IL-10、IL-17、IL-12、 IFN-γ、IFN-α、TNF-α.
CD4、CD8、CD4/CD8 | Day 0、day 7
  Flow cytometry will be used to detect serum CD4, CD8 and CD4/CD8 levels.
Vasoactive drugs applications | Day 0 to day 7
  The duration of vasoactive drug use will be recorded.
CRRT applications | Day 0 to day 7
  The duration of continuous renal replacement therapy will be recorded.
ECMO applications | Day 0 to day 7
  The duration of extracorporeal membrane oxygenation will be recorded.
All-cause mortality to day 28 | Up to 28 days
  The prognosis of patients on the 28th days will be counted.
All-cause mortality to day 60 | Up to 60 days
  The prognosis of patients on the 60th days will be counted.
ICU-free days | 2 year
  The prognosis of patients ICU length of stay will be counted.
Hospital-free days | 2 year
  The prognosis of patients total length of stay will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Lu, Doctor, Principal Investigator — Jiangsu Province Hospital of Traditional Chinese Medicine
Locations (1):
- Affiliated Hospital of Nanjing University of Chinese Medicine, Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No